CLINICAL TRIAL: NCT00479427
Title: A Double-blind, Placebo Controlled Cross-over Study of the Effects of the CB2 Compound of GW842166 in Patients With Osteoarthritis
Brief Title: A Study Of The Effects Of CB2 Compound Of GW842166 In Patients With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: CBA106191
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis pain assessments
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall study (Experimental): overall study population
  Interventions: Drug: GW842166; Drug: Placebo

INTERVENTIONS:
Drug: GW842166 — 100 mg once daily
Drug: Placebo — once daily

SUMMARY:
This is a double-blind, two-period, placebo controlled cross-over Phase IIa study. This study is to use CB2 compound of GW842166 in patients with osteoarthritis. The pain assessments and WOMAC questionnaires will be used in the study after the repeated dose to evaluate the efficacy of CB2 compound of GW842166.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 50 to 80 years of age.
* A female is eligible to participate in this study if she is of: a) non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal (more than 1 year since last menstrual cycle), had a tubal ligation or is surgical sterilised); or, b) child-bearing potential, has a negative pregnancy test (urine) at screen and baseline, and agrees to one of the following:

  * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; or
  * Implants of levonorgestral; or
  * Injectable progestogen; or
  * Oral contraception (combined or progestogen only); or
  * Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year; or
  * Barrier method only if used with any of the above acceptable methods.
* A diagnosis of primary osteoarthritis of the knee at least 3 months in symptom duration prior to screen. For patients with OA in both knees, an index knee will be specified.
* Meets American College of Rheumatology (ACR) criteria for symptomatic osteoarthritis of the knee as defined by knee pain and radiographic evidence of osteophytes (Altman 1986)
* Global functional status I, II or III according to ACR classification (see Appendix 5).
* Patient has a minimum of 40mm on the 100mm VAS (WOMAC pain subscale) at baseline / randomisation. In addition, baseline pain must be stable for at least 72 hours prior to randomisation based on patient's assessment.

Patient has a maximum of 80mm on the 100mm VAS (WOMAC pain subscale) at screening.

Exclusion Criteria:

* Intolerance of paracetamol.
* Any clinical or biological abnormality found at screening (other than those related to the disease under investigation) which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study (e.g. current malignancy, human immunodeficiency virus (HIV) infection, significant mental illness).
* QTc ≥450msecs based on a 12-lead ECG obtained over a brief recording period. This applies to QTc intervals measured either by Bazzett's or Fridericia's formula (machine or manual over-read, male or female subjects).
* Subjects with any one of creatinine, bilirubin, alanine aminotransferase (ALT) or aspartate aminotransfarase (AST) > 1.5 times the upper limit of normal (ULN) at screen are excluded. Subjects with two or more of bilirubin, ALT or AST above the ULN are excluded.
* Chronic Hepatitis B and C, as evidenced by positive Hepatitis B surface antigen (HbsAg) or Hepatitis C antibody
* History of chronic alcoholic liver disease
* Impaired renal function (estimated GFR<30mL/min)
* Use of potent CYP3A4 inhibitors (e.g. amiodarone, cyclosporine, diltiazem, elfinavir, indinavir, ritonavir, cimetidine, clarithromycin, erythromycin, fluconazole, itraconazole, ketoconazole, miconazole, nefazodone, verapamil)
* Use of methotrexate.
* Use of anticoagulants (warfarin, heparin) or anti-platelet aggregation agents (excluding low-dose aspirin) or a condition associated with decreased haemostasis
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* A history of clinically significant drug or alcohol abuse, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria [Hochberg, 1991]
* Participation in another investigational drug or device study during the 3 months prior to the Baseline/Randomisation Visit
* Inability or unwillingness to comply with study restrictions
* An unwillingness of male subjects to use a condom/spermicide, in addition to having their female partner use another form of contraception, such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if engaging in sexual intercourse with a female partner who could become pregnant. This criterion must be followed from the time of the first dose of study medication until three months after the last dose of study medication.

Exclusion criteria related to OA:

* Secondary causes of arthritis of the knee including septic arthritis, inflammatory joint disease, articular fracture, major dysplasias or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, and primary osteochondromatosis
* Had lower extremity surgery (including arthroscopy) within 6 months prior to screening or scheduled for surgery of any kind during the study period
* Significant prior injury to the index knee within 12 months prior to screen
* Use of lower extremity assistive devices other than a cane or knee brace (use of a 'shoe lift' is permitted)
* Disease of the spine or other lower extremity joints of sufficient degree to affect the index knee
* Any other musculoskeletal or arthritic condition that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study (i.e., currently symptomatic fractures or any concurrent rheumatic disease such as but not limited to fibromyalgia, rheumatoid arthritis, and Reiter's syndrome are excluded)
* Use of any analgesic, COX-2 inhibitor or NSAID [including topical NSAIDs; excluding low-dose aspirin (≤325mg per day)], other than protocol defined rescue therapy (paracetamol), within 5× half-life (in hours) prior to the first dosing day or during the study
* Corticosteroid use prior to baseline as follows:

  * Intra-articular injection of steroids to the index knee within the previous 3 months
  * Intra-articular steroid injections into any site other than the index knee within the
  * Intra-muscular corticosteroid injections within the previous 3 months
  * Oral corticosteroids within the previous 1 month
* Received hyaluronan injections into index knee within the previous six months prior to baseline
* Initiation of or change to an established physiotherapy program within 2 weeks prior to baseline or during the study period. An established physiotherapy program may be continued throughout the study period if unchanged in frequency and intensity Recent start or change in dose regimen (≤3 months prior to baseline) of any OA-specific therapies (i.e., nutraceutical products) including but not limited to chondroitin or keratin sulfate, s-adenosyl methionine (SAMe) and glucosamine preparations

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-07-06 (Actual); Primary Completion 2007-10-09 (Actual); Study Completion 2007-10-09 (Actual)

PRIMARY OUTCOMES:
Change in pain scores from Baseline to the end of treatment Western Ontario and McMasters University Osteoarthritis Index (WOMAC) using on the pain subscore for 6-8 weeks | Baseline (Day 1 pre-dose) and up to Day 14 of each treatment period (approximately up to 8 weeks)
  The index consisted of 24 questions (5 for pain, 2 for stiffness and 17 for physical and composite functions). The visual analog scale (VAS; 0-100 millimeter [mm]) was utilized in this study and participants were asked to rate joint pain they had in last 24 hours in the 5 pain items. Participants were asked to rate pain while performing following activities: walking on a flat surface, going up or down stairs; at night while in bed; sitting or lying and standing upright. Higher score (100) indicates extreme pain and lower score (0) indicates no pain. It was assessed on Day 1 pre-dose (Baseline), Day 1 (1 hour post-dose) and Day 14 (2-4 hours post-dose). Change from Baseline was planned to be calculated by subtracting Baseline value from post-Baseline value. Due to the early termination of this study, no formal statistical analysis was performed. Only summarized data is available.

SECONDARY OUTCOMES:
Quantitative Sensory Testing (QST) rating heat pain threshold and tolerance for 6-8 weeks | Up to Day 14 of each treatment period (approximately up to 8 weeks)
  Heat pain threshold was the temperature at which the participant first feels a painful stimulus. The heat pain threshold on normal skin was usually around 45 degree celcius. Mechanical pain threshold was assessed using an algometer to increase pressure against the skin of the affected joint until the point at which the participant reports pain. It was planned to assess for right knee and right forearm on Baseline (Day 1 pre-dose) and Day 14 (2-4 hours post-dose). Due to the early termination of this study, no formal statistical analysis was performed. Only summarized data is available.
Change from Baseline to the end of treatment in WOMAC stiffness subscore | Up to Day 14 of each treatment period (approximately up to 8 weeks)
  The participants were instructed to consider his/her response not only in terms of pain and functional impairment, but also in terms of consequences to his/her personal, conjugal, professional and social activities. The VAS; 0-100 (mm) was utilized in this study and participants were asked rate how much joint pain they have in last 24 hours in the 2 pain items. Participants were asked to rate pain while performing following activities: first awakening in the morning and sitting, lying or resting later in the day. Higher score (100) indicates extreme pain and lower score (0) indicates no pain. It was assessed on Baseline (Day 1 pre-dose) and Day 14 (2-4 hours post-dose). Change from Baseline was planned to be calculated by subtracting Baseline value from post-Baseline value. Due to the early termination of this study, no formal statistical analysis was performed. Only summarized data is available.
Change from baseline to the end of treatment in WOMAC physical function subscore | Baseline (Day 1 pre-dose) and up to Day 14 of each treatment period (approximately up to 8 weeks)
  The VAS; 0-100 (mm) was utilized in this study and participants were asked rate how much joint pain they have in last 24 hours in the 17 pain items. Participants were asked to rate pain while performing following activities: descending stairs; ascending stairs; rising from sitting; standing; bending to the floor; walking on a flat surface; getting in or out of a car/bus; going shopping; putting on your socks or tights; rising from bed; taking off your socks or tights; lying in bed; getting in or out of the bath; sitting; getting on or off the toilet; performing heavy domestic duties and performing light domestic duties. Higher score (100) indicates extreme pain and lower score (0) indicates no pain. It was assessed on Baseline (Day 1 pre-dose) and Day 14 (2-4 hours post-dose). Due to the early termination of this study, no formal statistical analysis was performed. Only summarized data is available.
Change from baseline to the end of treatment in participants' and Physician's Global assessment of arthritis condition | Baseline (Day 1 pre-dose) and up to Day 14 of each treatment period (approximately up to 8 weeks)
  The VAS; 0-100 (mm) was utilized in this study and participants were asked rate how much joint pain they have in last 24. Participants were asked 'considering all the ways your osteoarthritis (study knee) affects you (him/her), how are you doing today' by investigator for participants' (Physician's) Global assessment. Higher score (100) indicates very poor and lower score (0) indicates very well. It was assessed on Baseline (Day 1 pre-dose) and Day 14 (2-4 hours post-dose). Due to the early termination of this study, no formal statistical analysis was performed. Only summarized data is available.
Time for the 40 meter self-paced walk test and 11 step stair climb test | Up to Day 14 of each treatment period (approximately up to 8 weeks)
  The time taken for participant to walk for 40 meters from stationary to complete the walk and climb and descend 11 (dependent on site) steps with a handrail was recorded by the investigator or designee. The pain rate was also planned to assesse in participants by using 100 mm VAS after 40 meters walking. The pain was rated as 0 for No Pain and 100 for Extreme Pain. The time was also recorded for the participant to walk the first 20 meter in addition to the time for the complete walk. Due to the early termination of this study, this end point was not assessed.
Pain intensity (100mm VAS) for the 40 meter self-paced walk test and for 11 step stair climb test | Up to Day 14 of each treatment period (approximately up to 8 weeks)
  The VAS; 0-100 (mm) was utilized in this study and participants were asked to walk for 40 meters from stationary to complete the walk and climb and was recorded by the investigator or designee. Higher score (100) indicates extreme pain and lower score (0) indicates no pain. It was assessed on Baseline (Day 1 pre-dose) and Day 14 (2-4 hours post-dose). Due to the early termination of this study, this end point was not assessed.
Percentage of participants discontinuing due to lack of efficacy | Up to Day 14 of each treatment period (approximately up to 8 weeks)
  Due to the early termination of this study, this end point was not assessed.
Average total daily use of rescue medication | Up to Day 14 of each treatment period (approximately up to 8 weeks)
  Up to 3 grams of paracetamol in divided doses were allowed as rescue medication per day, but participants were advised that they must refrain from rescue medication within 24 hours prior to a clinic visit (Day 1 and 14). All rescue medication use was planned to be recorded in the diary card. Due to the early termination of this study, this end point was not assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom